CLINICAL TRIAL: NCT05873361
Title: Interest of Postoperative Follow-up of Asymptomatic Papillary Microcarcinomas on Patient Survival
Brief Title: Postoperative Follow-up of Asymptomatic Papillary Microcarcinomas on Patient Survival
Acronym: MIPTHYS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0059; 2023-A00294-41 (Other: ANSM)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Papillary Carcinoma
Keywords: Papillary Carcinoma; Postoperative; Follow-up
MeSH Terms: conditions — Carcinoma, Papillary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with a papillary microcarcinoma asymptomatic: Adult patients who have had a papillary microcarcinoma asymptomatic and who are followed.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire is about hypocalcemia, dysphonia and anxiety. It will be carried out by phone call for 10 minutes

SUMMARY:
This is a study assessing the interest of post-operative follow-up of asymptomatic papillary microcarcinomas. Today, this post-operative follow-up represents an economic cost and is a source of anxiety for patients.

The aim of this study is to determine the global survival of patients with asymptomatic papillary microcarcinoma to assess the interest of a post-operative ultrasound and/or biological follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uni or multifocal papillary microcarcinoma (cumulative size of foci <10mm) asymptomatic or not and who underwent partial or total thyroidectomy from 2012 to 2017.
* Non opposition patient
* Affiliation to a social security scheme

Exclusion Criteria:

* Lesion crossing the thyroid capsule, or cervical lymph node involvement clinical or histological cervical lymph node involvement.
* Patient under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with papillary microcarcinoma asymptomatic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Review of medical record

SECONDARY OUTCOMES:
Disease control rate | 10 years
  No recurrence clinically detected or by additional examen
Surgical complications rate | 10 years
  Dysphonia and hypocalcemia
Detection of recurrence rate | 10 years
  Recurrence detection by additional examen
Recovery surgical or iratherapie recovery rate | 10 years
  Anatomopathologic analysis
Anxiety evaluation | 1 month
  Likert scale
Prognostics survival criteria | 1 month
  Age during surgical

CONTACTS AND LOCATIONS:
Overall Officials: Agnès DUPRET-BORIES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France